CLINICAL TRIAL: NCT05331105
Title: A Multi-center, Open-label, Single-arm Phase II Study to Evaluate the Efficacy and Safety of HL-085 in the Treatment of Adult Participants With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas
Brief Title: HL-085 in Adults With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-106-II
Record Dates: First submitted 2022-03-15; First posted 2022-04-15 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibromas
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HL-085 (Experimental): HL-085 9mg BID
  Interventions: Drug: HL-085

INTERVENTIONS:
Drug: HL-085 — IIa: HL-085 capsule 9mg administered orally twice daily in a continuous 21-day treatment cycle. If required, dosing schedule can be adjusted to 12mg BID, 6mg BID, or other dosage regimens.
  IIb: HL-085 at the recommended dose or dosage regimen.

SUMMARY:
This is a Multi-center, Open-label, Single-arm Phase II Study to Evaluate the Efficacy and Safety of HL-085 in the treatment of Adult Participants with Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas(PN)

DETAILED DESCRIPTION:
The study includes 2 parts, phase IIa and IIb. Phase IIa is to evaluate the preliminary safety, pharmacokinetic characteristics and efficacy of HL-085, and to determine the recommended dose. To observe the 9mg dose level, approximately 15 patients will receive HL-085 at a dose of 9mg BID on a continuous dosing schedule(1 cycle=21 days). The investigator and sponsor will evaluate the safety and efficacy data to determine whether HL-085 9mg BID is appropriate. HL-085 12mg BID, 6mg BID, or other HL-085 dosing regimen will be observed as needed. A total of 15-35 patients will be enrolled in phase IIa. Phase IIb is to further evaluate the safety and efficacy of HL-085 in patients with NF1 and inoperable PN and is expected to enroll 35 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: patients must be ≥18 years of age at the time of study entry.
* Diagnosis: Patients must have inoperable and symptomatic plexiform neurofibromas(PN), and patients must have NF1 mutation or meet at least 1 of the following NF1 diagnostic criteria:

  ① ≥6 cafe-au-lait macules ;

  ② Axillary freckling or freckling in inguinal regions;

  ③ ≥2 Lisch nodules (iris hamartomas);

  ④ A distinctive bony lesion such as dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex);

  ⑤ An optic pathway glioma;

  ⑥ First-degree relative with NF1.
* Patients must have a measurable lesion, defined as at least 3 cm in length, amenable to MRI for efficacy assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients are able to understand and voluntarily sign a written informed consent form.
* Patients must be willing and able to complete study procedures and follow-up examinations.

Exclusion Criteria:

* Patients who are unable to undergo MRI scans (prosthesis, prosthesis, braces, etc.) or patients with lesions that cannot be evaluated by MRI.
* Patients do not have adequate organ function.
* Patients who are unable to take drugs orally, have difficulty swallowing or anything that may lead to inadequate drug absorption.
* Prior treatment with MEK 1/2 inhibitors.
* Patients known to be allergic to the ingredients or analogues of the study drug.
* Patients with previous or current retinal diseases such as retinal vein occlusion (RVO), retinal pigment epithelium detachment (RPED), central serous retinopathy (CSR), etc. (except retinopathy caused by research diseases).
* With infections or other uncontrolled disease.
* Strong CYP2C9 inhibitors or inducers within 7 days before treatment of the study drug.
* Patients who received surgery within 4 weeks or radiotherapy within 6 weeks before enrollment.
* Patients who participated in any other clinical study treatment within 4 weeks before enrollment.
* Patients treated with anti-NF1 treatment with unresolved chronic toxicity.
* Clinical judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end of cycle 4,8,12,16,20,24,28,32.Then after every 8 cycles(each cycle is 21 days)
  To assess the efficacy of HL-085 on the tumor volume (plexiform neurofibromas) using volumetric MRI per REiNS criteria. ORR is defined as the percentage of patients who have achieved a confirmed Partial Responses (PR) or Complete Responses (CR).

SECONDARY OUTCOMES:
Disease Control Rate（DCR） | At the end of cycle 4,8,12,16,20,24,28,32.Then after every 8 cycles(each cycle is 21 days)
  Defined as the percentage of patients who have achieved a confirmed response of CR or PR or SD
Duration of Overall Response（DOR） | At the end of cycle 4,8,12,16,20,24,28,32.Then after every 8 cycles(each cycle is 21 days)
  Defined as the time from first achieved CR or PR to disease progression
Progression Free survival (PFS) | From date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Defined as the time from first dosing (C1D1) to date of first observed progression or death from any cause (whichever comes first)
Pharmacokinetic characteristics | During the intervention
  AUC

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Chair — Shanghai Kechow Pharma, Inc.
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided